CLINICAL TRIAL: NCT01748695
Title: A Phase IIa, Randomized, Double-blind, Placebo-controlled, Two-period Cross-over Study Evaluating the Safety, Tolerability and Efficacy of V158866 in Central Neuropathic Pain Following Spinal Cord Injury
Brief Title: A Safety, Tolerability and Efficacy Study of V158866 in Central Neuropathic Pain Following Spinal Cord Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Vernalis (R&D) Ltd (Industry)
Responsible Party: Principal Investigator, Christine N. Sang, MD, MPH, Dr Christine Sang, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: V158866-2Pa-01
Record Dates: First submitted 2012-12-11; First posted 2012-12-12 (Estimated); Results first posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Neuropathic Pain Due to Spinal Cord Injury
Keywords: Neuropathic pain; Spinal cord injury
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo followed by V158866 (Experimental): Placebo once per day for 4 weeks followed by V158866 450mg once per day for 4 weeks
  Interventions: Drug: V158866; Drug: Placebo
- V158866 followed by Placebo (Experimental): V158866 450mg once per day for 4 Weeks followed by Placebo once per day for 4 Weeks
  Interventions: Drug: V158866; Drug: Placebo

INTERVENTIONS:
Drug: V158866
Drug: Placebo

SUMMARY:
The purpose of this study is to investigate whether V158866 is safe and effective for the treatment of neuropathic pain due to spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 - 65 years
* documented spinal cord injury at or below T5
* moderate pain at or below the level of the spinal cord injury for at least 3 months
* compliant with daily diary
* stable pain scores on the NRS
* mean pain intensity of at least 4 and not more than 9 on the NRS (or if the mean NRS score is >9, the mean Gracely score must be ≤19)

Exclusion Criteria:

* women of child-bearing potential
* men who intend to father a child
* a history of multiple drug allergies, hypersensitivity to any cannabinoid
* an increased risk of seizure
* evidence of depression and/or a score of >19 on the BDI-II
* suicidal ideation or suicidal behavior in the past 10 years
* a history of substance abuse or dependence within the past year, excluding nicotine and caffeine
* a positive urine test for cannabis at screening
* taking excluded medications that cannot be stopped
* a positive pregnancy test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine N Sang, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Translational Pain Research, Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Included a 14-day period to exclude non-compliers, extremes of pain ratings, and those with high variability
Period: First Intervention (4 Weeks)
Arm/Group | Placebo Followed by V158866 | V158866 Followed by Placebo
Started | 14 | 11
Completed | 14 | 11
Not Completed | 0 | 0
Period: Second Intervention (4 Weeks)
Arm/Group | Placebo Followed by V158866 | V158866 Followed by Placebo
Started | 14 | 11
Completed | 14 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- V158866 and Placebo: Placebo once per day for 4 weeks followed by V158866 450mg once per day for 4 weeks or vice versa
Arm/Group | V158866 and Placebo
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 18

OUTCOME MEASURES:

1. Primary Outcome: Mean Pain Intensity (NRS)
Description: Numerical Rating Scale, measuring the intensity of pain from 0 to 10, with 0 being no pain and 10 being worst pain imaginable. The comparison of the overall pain intensity, calculated as the mean of the last 7 days on treatment, for each treatment period (V158866 compared to placebo).
Time Frame: 4 Weeks
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo: Placebo once per day for 4 weeks
- V158866: V158866 450mg once per day for 4 weeks
Arm/Group | Placebo | V158866
Number analyzed (Participants) | 25 | 25
units on a scale | 5.93 (0.148) | 5.89 (0.148)
Statistical Analysis 1: Comparison: Placebo vs V158866; Test type: Superiority or Other; p = 0.834, Regression, Linear — Based on a linear mixed measures model with treatment and period included as fixed effects, subject included as a random effect and between- and within- subject baseline covariates included

2. Primary Outcome: Safety and Tolerability of V158866 Compared to Placebo
Description: Safety and tolerability were measured by occurrence of treatment-emergent adverse events; data represents the number of subjects who experienced treatment-emergent adverse events during each treatment period.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | V158866
Number analyzed (Participants) | 25 | 25
Participants | 7 | 12

ADVERSE EVENTS:
Time Frame: From start of study participation until all adverse events had resolved following study participation, an average of 4 months
Description: All events that were possibly, probably, or definitely related to study medication
Arm/Group | Placebo | V158866
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 7/25 | 12/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | V158866 (N=25)
Difficulty Concentrating (Nervous system disorders) | 0 (0) | 3 (3)
Fatigue (Sleepiness) (Nervous system disorders) | 0 (0) | 4 (4)
Headache (Nervous system disorders) | 6 (6) | 2 (2)
Drowsiness (Nervous system disorders) | 2 (2) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No